CLINICAL TRIAL: NCT03750825
Title: Are Smokers Switching to Vaping at Lower Risk for Cancer?
Brief Title: Are Smokers Switching to Vaping at Lower Risk for Cancer? (Electronic Cigarettes and Cancer Risk)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California (Other)
Responsible Party: Principal Investigator, Ahmad Besaratinia, Professor, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS-18-00744
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cigarette Smoking
Keywords: Electronic Nicotine Delivery System
MeSH Terms: conditions — Cigarette Smoking; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Vapers (Experimental): Smokers will switch to NIDA Standard Research E-cigarette (SREC).
  Interventions: Device: NIDA Standard Research E-cigarette (SREC)
- Smokers (No Intervention): Smokers will continue to smoke.
- Nonsmokers non-vapers (No Intervention): Control nonsmokers non-vapers will continue to refrain from smoking or vaping.

INTERVENTIONS:
Device: NIDA Standard Research E-cigarette (SREC) — Smokers will switch to NIDA Standard Research E-cigarette (SREC).
  Arms: Vapers

SUMMARY:
This project will address a growing public health concern, namely, the health risks or benefits of e-cig use relative to cigarette smoking. The investigators will use biomarkers of early effects of relevance to cancer to determine the carcinogenic potential of e-cig use relative to cigarette smoking in oral epithelium, which is a target tissue for smoking-associated cancer. The study population will consist of one group of smokers who are interested in switching to e-cig use (Grp 1), one group of smokers who do not intend to change their smoking habits (Grp 2), and one group of non-users who would like to maintain their nonsmoking non-vaping status (Grp 3); The total number of participants in this project is 150 (n = 50, each group). The investigators will use an integrative 'multi-omics' approach complemented with single-locus/gene validation analyses to detect temporal changes in the genome, epigenome, and transcriptome relevant to cancer in the oral cells of the participants as the intervention progresses.

DETAILED DESCRIPTION:
Electronic cigarettes (e-cig) are increasingly popular among adult smokers and adolescent never smokers. Chemical analyses of e-cig vapor and liquid have shown the presence of many of the same carcinogens as those found in cigarette smoke, albeit in generally lower concentrations. However, the carcinogenic potential of e-cig has not been investigated in e-cig users (otherwise known as 'vapers'). The investigators will investigate the cancer-causing potential of e-cig use as compared to cigarette smoking by quantifying molecular changes linked to risk of cancer in smokers who switch to e-cig use vs. those who maintain their smoking habits. Leveraging a source population for ongoing studies on e-cig, the investigators will recruit smokers who are interested in switching to e-cig use, and two control groups of non-vapers, including smokers and nonsmokers who do not intend to change their smoking and nonsmoking status, respectively (n = 50, each group). Smokers consenting to switch completely to e-cig will be assigned to a 3-month intervention with a standard e-cig with fully described product characteristics. Control groups will maintain their smoking/nonsmoking habits during the intervention. At weekly intervals, the investigators will verify participants' compliance through personal interviews, CO breath tests, cotinine quantification, and vaping/smoking topography measurements. The investigators will use a non-invasive brushing technique to collect oral cells from the inside of the cheeks of all participants at baseline and every 2 weeks, afterwards. The investigators will use an integrative 'multi-omics' approach complemented with single-locus/gene validation analyses to detect temporal changes in the genome, epigenome, and transcriptome relevant to cancer in the oral cells of the participants as the intervention progresses.

ELIGIBILITY:
Inclusion Criteria:

* Being male or female between the ages of 22-55;
* Being able to read and write in English and understand and give informed consent;
* Giving consent to strictly follow the study protocol throughout the study;
* Not planning to move, take an extended vacation, or undergo surgery during the study;
* Reporting smoking of > 5 manufactured cigarettes per day for at least 1 year (applicable to participants who will undergo intervention with e-cig (Grp 1) or continue to smoke (Grp 2) only); and
* Presenting with an expired air CO measurement of > 7 parts per million (ppm) at baseline (applicable to participants who will undergo intervention with e-cig (Grp 1) or continue to smoke (Grp 2) only).

Exclusion Criteria:

* Having oral infection/inflammation, gum disease, dental decay, immune system disorders, diabetes, respiratory diseases (e.g., asthma), or kidney diseases;
* Having any unstable or significant medical condition (e.g., symptomatic heart conditions) in the past 12 months ;
* Having body mass index < 18 kg/m2 or > 40 kg/m2
* Being pregnant or having a baby in the past 12 months;
* Having uncontrolled mental illness or substance abuse (e.g., alcoholism) or inpatient treatment for those conditions in the past 12 months;
* Having used recreational or illicit drugs in the past 3 months;
* Having used any medication known to induce/inhibit CYP450 2A6 enzyme;
* Having any known allergy to propylene glycol/vegetable glycerin (applicable participants who will undergo intervention with e-cig (Grp 1) only); and
* Having another member of household participating in the study.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Genetic changes | 3 months
  Number and location of DNA damage
Epigenetic changes | 3 months
  Number of epigenetic marks

SECONDARY OUTCOMES:
Gene expression | Every 2 weeks for 3 months
  Relative gene expression
DNA methylation | Every 2 weeks for 3 months
  Pattern and distribution of aberrant DNA methylation
Histone modifications | Every 2 weeks for 3 months
  Pattern and distribution of histone marks
Mutation | Every 2 weeks for 3 months
  Frequency and location of mutations

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Besaratinia, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Health Sciences Campus, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.